CLINICAL TRIAL: NCT03699930
Title: Impact of Neuromodulation on Language Impairments in Stroke Patients: a Multimodal Double-blind Randomized Controlled Study
Brief Title: Impact of Neuromodulation on Language Impairments in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Casa Colina Hospital and Centers for Healthcare (Other)
Responsible Party: Principal Investigator, Amy Zheng, Research Scientist, Casa Colina Hospital and Centers for Healthcare
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TDCS
Record Dates: First submitted 2018-07-27; First posted 2018-10-09 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Stroke; Aphasia
Keywords: transcranial direct current stimulation; stroke; aphasia; speech therapy; neurorehabilitation; neuromodulation; language function; neuroplasticity; neuroimaging; EEG; MRI; genetics; language disorders
MeSH Terms: conditions — Stroke; Aphasia; Communication Disorders; Language; Language Disorders | interventions — Transcranial Direct Current Stimulation; Speech Therapy

STUDY DESIGN:
Intervention Model Description: double-blind quasi-randomized controlled design
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The only person knowing about this assignment will be the Principal Investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- tDCS + speech therapy (Active Comparator): Participants will receive 20 minutes of anodal tDCS paired with speech and language therapy over five consecutive days.
  Interventions: Device: tDCS; Behavioral: Speech and language therapy
- sham + speech therapy (Sham Comparator): Participants will receive 20 minutes of sham tDCS paired with speech and language therapy over five consecutive days.
  Interventions: Device: tDCS; Behavioral: Speech and language therapy

INTERVENTIONS:
Device: tDCS — Anodal or sham tDCS will be applied to the scalp.
Behavioral: Speech and language therapy — A trained speech pathologist will administer the speech and language therapy.

SUMMARY:
Up to 40% of stroke survivors suffer from aphasia, making recovery of language abilities a top priority in stroke rehabilitation. Conventional speech and language therapy may have limited effectiveness. Leveraging multimodal data (behavioral, neuroimaging, and genetics), this study aims to 1) evaluate the efficacy of combining tDCS with speech therapy, 2) examine neural changes associated with recovery, 3) identify factors influencing response to treatment.

DETAILED DESCRIPTION:
Approximately one million people in the United States are living with aphasia, an acquired neurological disorder affecting the ability to use and/or understand language. This communication impairment affects up to 40% of stroke patients. Stroke victims usually prioritize speaking, writing, and walking as the three most important rehabilitation goals, two of these goals therefore involving communication. Conventional speech therapy strategies have nevertheless limited effectiveness in post-stroke aphasia. Indeed, approximately half of those affected will remain in this state despite intensive speech therapy. Effective novel treatment is therefore warranted to improve recovery in these patients. Recent evidence suggests that transcranial direct current stimulation (tDCS), a non-invasive, low-cost neuromodulation technique, applied in conjunction with speech therapy may be more effective in promoting language recovery than behavioral intervention alone.

A double-blind quasi-randomized controlled study will be carried out in chronic post-stroke aphasics. Participants will be assigned to either the tDCS group or to the sham (placebo) group and will receive 20 minutes of concurrent speech and language therapy by a trained speech therapist over five consecutive days. Behavioral, EEG, and MRI data will be acquired within one week before and after intervention. Genetic samples will be collected once. Secondary behavioral outcome measures will be performed again 3 months following tDCS/sham intervention to assess long-term benefits.

ELIGIBILITY:
Inclusion Criteria:

* Between ages 18-85
* At least 12 months post stroke
* Diagnosed with aphasia due to ischemic or hemorrhagic stroke
* English speaking
* Right handed prior to stroke

Exclusion Criteria:

* Nonverbal
* Other neurological diseases/disorders
* Not MRI-compatible (e.g. claustrophobia, metal implants in the head)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Change in Western Aphasia Battery-Revised scores | At baseline and at week 3
  WAB-R is an instrument for assessing the language function of adults with suspected neurological disorders as a result of a stroke.

SECONDARY OUTCOMES:
Change in Magnetic Resonance Imaging (MRI) | At baseline and at week 3
  MRI scans will be acquired on a Siemens Magnetom Verio 3T Scanner at Casa Colina Imaging Center to assess structural changes.
Change in resting state Electroencephalograph (EEG) signals | At baseline and at week 3
  Using a B-Alert wireless EEG system, we will perform eyes-open resting-state EEG recordings to assess power spectral density changes.
Change in Test of Nonverbal Intelligence (TONI-4) | At baseline and at week 3
  TONI-4 is a language-free intelligence test for evaluating those with limited language ability.
Change in Communication Outcomes after Stroke (COAST) | At baseline, at week 3, and at week 17
  The COAST is used to assess self-perceived communication effectiveness for people with aphasia.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) | At baseline, at week 3, and at week 17
  PROMIS is used to assess physical, mental, and social health.
Change in Stroke and Aphasia Quality of Life Scale-39 (SAQOL-39) | At baseline, at week 3, and at week 17
  The SAQOL-39 is used to assess health-related quality of life in people with long-term aphasia.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Zheng, PhD, Principal Investigator — Casa Colina Hospital and Centers for Healthcare
Locations (1):
- Casa Colina Hospital and Centers for Healthcare, Pomona, California, United States

REFERENCES:
- [Derived] Zheng ZS, Wang J, Lee S, Wang KX, Zhang B, Howard M, Rosario E, Schnakers C. Cerebellar transcranial direct current stimulation improves quality of life in individuals with chronic poststroke aphasia. Sci Rep. 2025 Feb 26;15(1):6898. doi: 10.1038/s41598-025-90927-y. PMID 40011597